CLINICAL TRIAL: NCT03683940
Title: A Prospective Pilot Study of Lung Cancer Screening in Patients at High Risk for Lung Cancer Who Do Not Meet Current Screening Guidelines
Brief Title: Pilot Study of High Risk Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15-1694.cc
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: Pilot Study; High Risk; Prospective; Screening
MeSH Terms: conditions — Lung Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Other): Subjects will undergo a low dose non contrast CT chest for lung cancer screening.
  Interventions: Diagnostic Test: Screening

INTERVENTIONS:
Diagnostic Test: Screening — Subjects will undergo a low dose non contrast CT chest for lung cancer screening. The test will be performed by the UCH Radiology Department and read by board-certified chest radiologists using Lung-RADS criteria.

SUMMARY:
This study is a prospective trial of 200 individuals at high risk for lung cancer who are not eligible for lung cancer screening under current screening guidelines.

DETAILED DESCRIPTION:
This study is a prospective trial of 200 individuals at high risk for lung cancer who are not eligible for lung cancer screening under current screening guidelines. Potential subject's 6 yr lung cancer risk must exceed 1.5% by the Tammamagi PLCO2012m calculator. Patients will undergo a non contrast CT chest for lung cancer screening. This cutoff should encompass in excess of 80% of all lung cancer cases (10). However, in patients 78-82 years old we will set the 6 yr lung cancer risk threshold at 4.0% as these patients will typically have other competing risks of death and this may potentially limit screening benefit in these older individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 40-82 yrs of age.
2. Presenting for lung cancer screening evaluation.
3. Calculated 6 yr lung cancer risk >1.5% for patients 40-77 years of age or >4% for patients 78-82 years of age.
4. Able and willing to provide informed consent.

Exclusion Criteria:

1. Eligible for clinically indicated lung cancer screening (55-80 yr old, >30 pky smoking history, still smoking or quit smoking within the last 15 yr).
2. Chest CT performed within the last year.
3. Life expectancy less than 6 months.
4. Symptoms clinically consistent with lung cancer.
5. Unable or unwilling to undergo treatment for lung cancer.
6. Any individual who does not give oral and written consent for participation.

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Lung Cancer Screening | Duration of the study, up to 3 years
  Prospectively identify patients for lung cancer screening using risk calculators
Medical Outcomes | Duration of the study, up to 3 years
  Evaluate health outcomes of CT screening by assessing the number and stage of lung cancers detected by screening using Lung-RADS criteria
Medical Outcomes | Duration of the study, up to 3 years
  Evaluate health outcomes of CT screening by assessing the number and stage the spectrum of other radiographic abnormalities detected using Lung-RADS criteria
Economic Outcomes | Duration of the study, up to 3 years
  Evaluate the costs associated with managing lung cancers detected by screening
Economic Outcomes | Duration of the study, up to 3 years
  Evaluate the costs associated with managing the spectrum of other radiographic abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Melissa New, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

REFERENCES:
- [Derived] Hirsch EA, New ML, Brown SL, Malkoski SP. Results of a pilot risk-based lung cancer screening study: outcomes and comparisons to a Medicare eligible cohort. Discov Oncol. 2023 Aug 29;14(1):160. doi: 10.1007/s12672-023-00773-5. PMID 37642787

DOCUMENTS (1):
  • Informed Consent Form (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03683940/ICF_000.pdf